CLINICAL TRIAL: NCT04377945
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Part Study in Parkinson's Disease Patients With Dyskinesia to Assess the Efficacy and Safety/Tolerability of Fixed Dose Combinations of JM-010 and Its Individual Components
Brief Title: Study in Parkinson's Disease Patients With Dyskinesia With Combinations of JM-010 and Its Individual Components
Acronym: SHINE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK-JM-201
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Dyskinesias; Parkinson Disease
MeSH Terms: conditions — Dyskinesias; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1, JM-010 component Group A (Experimental): Part 1, JM-010 component Group A
  Interventions: Drug: Part 1, JM-010 component Group A
- Part 1, JM-010 component Group B (Experimental): Part 1, JM-010 component Group B
  Interventions: Drug: Part 1, JM-010 component Group B
- Part 1, JM-010 component Group C (Experimental): Part 1, JM-010 component Group C
  Interventions: Drug: Part 1, JM-010 component Group C
- Part 1, Placebo Group (Placebo Comparator): Part 1, Placebo Group
  Interventions: Drug: Part 1, Placebo Group
- Part 2, JM-010 combination Group A (Experimental): Part 2, JM-010 combination Group A
  Interventions: Drug: Part 2, JM-010 combination Group A
- Part 2, JM-010 combination Group B (Experimental): Part 2, JM-010 combination Group B
  Interventions: Drug: Part 2, JM-010 combination Group B
- Part 2, JM-010 component Group C (Experimental): Part 2, JM-010 component Group C
  Interventions: Drug: Part 2, JM-010 component Group C
- Part 2, Placebo Group (Placebo Comparator): Part 2, Placebo Group
  Interventions: Drug: Part 2, Placebo Group

INTERVENTIONS:
Drug: Part 1, JM-010 component Group A — JM-010 component Group A
  Arms: Part 1, JM-010 component Group A
Drug: Part 1, JM-010 component Group B — JM-010 component Group B
  Arms: Part 1, JM-010 component Group B
Drug: Part 1, JM-010 component Group C — JM-010 component Group C
  Arms: Part 1, JM-010 component Group C
Drug: Part 1, Placebo Group — Placebo Group
  Arms: Part 1, Placebo Group
Drug: Part 2, JM-010 combination Group A — JM-010 combination Group A
  Arms: Part 2, JM-010 combination Group A
Drug: Part 2, JM-010 combination Group B — JM-010 combination Group B
  Arms: Part 2, JM-010 combination Group B
Drug: Part 2, JM-010 component Group C — JM-010 component Group C
  Arms: Part 2, JM-010 component Group C
Drug: Part 2, Placebo Group — Placebo Group
  Arms: Part 2, Placebo Group

SUMMARY:
This is a two-part, double-blind, placebo-controlled, randomized, multicenter Phase 2 clinical trial of JM-010 in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
This is a two-part, Phase 2, double-blind, placebo-controlled, randomized, multicentre study.

Subjects with a diagnosis of PD and dyskinesias in PD will complete a Screening Visit to assess eligibility to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Is able to read, understand, and provide written, dated informed consent prior to Screening Visit.
* Is male or female, between 18 and 85 years of age at Screening Visit.
* Is diagnosed with idiopathic PD that meets UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* Has experienced dyskinesia
* Has stable peak-effect dyskinesia
* Has more than one hour of "ON" time with troublesome dyskinesia

Exclusion Criteria:

* Has undergone surgery for the treatment of PD
* Has a current diagnosis of Substance Use
* Has psychiatric diagnosis of acute psychotic disorder or other psychiatric diagnoses
* Has current seizure disorders requiring treatment with anticonvulsants.

Other criteria related to other medical conditions to be referred to the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | Week 12
  Unified Dyskinesia Rating Scale (Scoring range: 0-104), higher score indicates more severe dyskinesia

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Week 12
  Movement Disorder Society Unified Parkinson's Disease Rating Scale (Part III Scoring range: 0-137), higher score indicates more severe motor impairment

CONTACTS AND LOCATIONS:
Overall Officials: Sooyeon Park, Study Director — Bukwang Pharmaceutical
Locations (2):
- United States (2):
  - Bukwang Investigator site, Miami, Florida
  - Bukwang Investigator site, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No